CLINICAL TRIAL: NCT01590121
Title: A Questionnaire Based Study to Evaluate the Safety of Flying in Hereditary Haemorrhagic Telangiectasia (HHT)
Brief Title: Hereditary Haemorrhagic Telangiectasia Flight Safety Study
Acronym: Flying and HHT
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CLS/20
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: Previous flight by aeroplane
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pateints with hereditary haemorrhagic telangiectasia
  Interventions: Other: Aeroplane flight in the past- no active intervention for study; Other: Questionnaire

INTERVENTIONS:
Other: Aeroplane flight in the past- no active intervention for study — Aeroplane flight(s) previously taken by study participants
Other: Questionnaire — Flight by aeroplane (previous)

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT) is a condition in which sufferers have abnormal blood vessels which makes them more likely to bleed than other people, particularly in the lungs, which results in low blood oxygen levels. Flying may make this worse and cause problems. The investigators want to know if there are an increased number of problems on flights compared to on land.

The investigators currently do not have any evidence based guidelines on air travel to best advice people who suffer with HHT. The investigators would therefore like to ask individuals who have HHT about their experience on a flight, using a postal questionnaire.

DETAILED DESCRIPTION:
Individuals with Hereditary Haemorrhagic Telangiectasia (HHT) previously reviewed at HHTIC London will be sent an invitation to participate in a short questionnaire study.

Quantitative variables from the questionnaires for statistical analysis will be the number of individuals responding (and number of questionnaires sent out); number of flights taken and number of complications, subgrouped by type, and flight duration in hours. Complication rates will be expressed as proportion of person flight hours.

The quantitative data from the questionnaire will then be compared with quantitative data from patients' medical records using non parametric methods such as Mann Whitney for univariate analyses.

ELIGIBILITY:
Inclusion Criteria:

HHT

Exclusion Criteria:

Unable to provide informed consent

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HHT patients previously assesses at Hammersmith Hospital, England
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD MA MB BChir FRCP, Principal Investigator — Imperial College London
Locations (1):
- HammersmithHospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mason CG, Shovlin CL. Flight-related complications are infrequent in patients with hereditary haemorrhagic telangiectasia/pulmonary arteriovenous malformations, despite low oxygen saturations and anaemia. Thorax. 2012 Jan;67(1):80-1. doi: 10.1136/thoraxjnl-2011-201027. Epub 2011 Sep 26. PMID 21953065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pateints With Hereditary Haemorrhagic Telangiectasia
Started | 156
Completed | 156
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pateints With Hereditary Haemorrhagic Telangiectasia
Number analyzed (Participants) | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 53
Age, Continuous [Mean (Full Range); unit: years] | 55 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 156

OUTCOME MEASURES:

1. Primary Outcome: HHT Patients Who by the Questionnaire Did or Did Not Self Report a Medical Complication During Flight
Description: Of all patients who were sent the questionnaire, this comparison was limited to those who had taken a flight, either long haul or short haul.
  Participants were compared as to whether they did or did not suffer a flight complication.
Time Frame: Patient were asked to report all flights taken up until questionnaire completion aged 18-90 (mean 55)ys. 145 HHT-affected respondents had flown for 18,943 hours over 3,950 flights.
Population: Percentage of individuals who reported complications
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- HHT Flight Group: Study participants who self reported by questionnaire that they took one or more flights by aeroplane.
  We excluded two patients who had flown extensively due to their occupation, reporting over 10,000 flights between them (pilot and cabin crew) as this was a self-selecting group who would substantially skew the data.
Arm/Group | HHT Flight Group
Number analyzed (Participants) | 145
percentage of patients | 77 [69.6 to 83.5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Pateints With Hereditary Haemorrhagic Telangiectasia
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156
Other Adverse Events (participants affected / at risk) | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes